CLINICAL TRIAL: NCT01069614
Title: A Skin Stretching Wound Closure System
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Moris Topaz, MD, PhD, Hillel Yaffe Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-09
Record Dates: First submitted 2010-02-07; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Wounds; Injuries
Keywords: Equipment and supplies
MeSH Terms: conditions — Wounds and Injuries

ARMS (1):
- Skin stretching device (Experimental): Skin stretching device
  Interventions: Device: TopClosure 3S System

INTERVENTIONS:
Device: TopClosure 3S System

SUMMARY:
A skin stretching device has been designed to stretch tissue prior to surgery, during surgery and in order to secure wounds following surgery. The device may be used in non-invasive and invasive applications.

ELIGIBILITY:
Inclusion Criteria:

* Hard to close wounds

Exclusion Criteria:

* Non-cooperative patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of wound closure

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel